CLINICAL TRIAL: NCT01086254
Title: Randomized Phase 2 Study of Gemcitabine/Cisplatin With or Without SAR240550 (BSI-201), a PARP1 Inhibitor, in Patients With Stage IV Non-small Cell Lung Cancer
Brief Title: SAR240550 in Combination With Gemcitabine/Cisplatin in Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCD11420; 2009-017270-21 (EudraCT Number); U1111-1116-5404 (Other: UTN)
Record Dates: First submitted 2010-03-11; First posted 2010-03-15 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Non-small Cell Lung Cancer Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — iniparib; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iniparib/ Gemcitabine/ Cisplatin (Experimental): Iniparib, 5.6 mg/kg, 60-min IV infusion twice weekly (days 1, 4, 8, and 11). Infusion starts after completion of GC regimen administration.
  Gemcitabine, 1250 mg/m2, 30-min IV infusion on day 1 and day 8 and cisplatin 75mg/m², 3- to 4-hour IV infusion on day 1 of each 3-week cycle after the end of gemcitabine infusion.
  Interventions: Drug: Iniparib; Drug: gemcitabine; Drug: cisplatin
- Gemcitabine/ Cisplatin (Active Comparator): Gemcitabine, 1250 mg/m2, 30-min IV infusion on day 1 and day 8 and cisplatin 75mg/m², 3- to 4-hour IV infusion on day 1 of each 3-week cycle after the end of gemcitabine infusion.
  Interventions: Drug: gemcitabine; Drug: cisplatin

INTERVENTIONS:
Drug: Iniparib — Pharmaceutical form: solution for infusion
  Route of administration: 60-minute IV infusion
  Other Names: SAR240550; BSI-201
  Arms: Iniparib/ Gemcitabine/ Cisplatin
Drug: gemcitabine — Pharmaceutical form: solution for infusion
  Route of administration: 30-minute IV infusion
Drug: cisplatin — Pharmaceutical form: solution for infusion
  Route of administration: 1- to 4-hour IV infusion, according to the local standard

SUMMARY:
Primary Objective:

* to assess the objective response rate (ORR) of Iniparib (SAR240550) administered as a 60-min intravenous infusion twice weekly, when combined to gemcitabine/cisplatin chemotherapy regimen (GCS) as well as with the standard regimen of gemcitabine/cisplatin (GC) in patients with stage IV non small cell lung cancer.

Secondary objectives are:

* to assess the safety profiles of the study combination GCS and of the standard regimen GC;
* to assess the progression free survival and the overall survival in both arms;
* to assess the relationship between DNA repair pathway characteristics of tumors at baseline and clinical outcome of disease.
* to assess the effect of Iniparib on PAR level in peripheral blood mononuclear cells (PBMC). (As of 10 September 2010, the collection of PBMC is temporarily discontinued.)

DETAILED DESCRIPTION:
The duration of the study for a patient will include a period for inclusion of up to 3 weeks. The patients may continue treatment up to a maximum of 6 cycles or until disease progression, unacceptable toxicity or consent withdrawal, followed by a minimum of 30-day follow-up after the last study treatment administration.

Patients will be followed for at least 30 days after the last administration of study treatment for safety purpose. In case of study treatment discontinuation without disease progression, efficacy data will be collected every 6 weeks until disease progression, death or end of study whatever comes first. After disease progression, the patient will be followed-up every 12 weeks (3 months) for overall survival (OS) until death or end of study whatever comes first.

The end of the study will be one year after the first dose of the last treated patient.

ELIGIBILITY:
Inclusion criteria:

* Stage IV disease (including stage IIIB with pleural effusion) with no prior systemic therapy. Adjuvant therapy is allowed if ended more than 1 year before inclusion in the study.
* Histologically confirmed squamous cell bronchogenic carcinoma OR non squamous cell carcinoma.
* Patients with previous radiotherapy as definitive therapy for locally advanced non-small cell lung cancer are eligible, as long as the selected measurable lesions are outside the original radiation therapy port. Radiation therapy must have been completed >4 weeks prior to study entry.
* Palliative radiotherapy must have been completed > 2 weeks prior to study entry. Irradiated lesions may not serve as measurable lesions.
* At least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Adequate bone marrow reserve.
* Adequate liver and renal function.
* Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to start of treatment.

Exclusion criteria:

* Prior treatment with gemcitabine, platinum salts or any PARP inhibitor class compound.
* Past or current history of neoplasm other than the entry diagnosis, with the exception of treated non-melanoma skin cancer or carcinoma in-situ of the cervix, or other cancers cured by local therapy alone and with an expected disease-free survival of > or = 5 years.
* Major medical conditions that might affect study participation e.g. cardiac disease, uncontrolled infection (>Grade 2).
* Presence of active brain metastases.
* A major surgical procedure, open biopsy, or significant traumatic injury within 28 days of beginning treatment, or anticipation of the need for major surgery during the course of the study.
* Any history of medical or psychiatric condition or laboratory abnormality that, in the opinion of the investigator, may increase the risks associated with the study participation or administration of the investigational products, or that may interfere with the interpretation of the results
* Grade 2 or higher ear and labyrinth disorders.
* Known or suspected allergy/hypersensitivity to any agent given in the course of this trial.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
overall response rate (ORR) that is defined in the RECIST 1.1 version, as: complete response rate + partial response rate | up to a maximum follow-up of 25 weeks

SECONDARY OUTCOMES:
progression free survival | up to a maximum of 2 years
overall survival | up to a maximum of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (14):
- France (4):
  - Sanofi-Aventis Investigational Site Number 250002, Caen
  - Sanofi-Aventis Investigational Site Number 250003, Marseille
  - Sanofi-Aventis Investigational Site Number 250004, Toulouse
  - Sanofi-Aventis Investigational Site Number 250001, Villejuif
- Germany (3):
  - Sanofi-Aventis Investigational Site Number 276003, Essen
  - Sanofi-Aventis Investigational Site Number 276002, Gauting
  - Sanofi-Aventis Investigational Site Number 276001, Großhansdorf
- Italy (3):
  - Sanofi-Aventis Investigational Site Number 380003, Livorno
  - Sanofi-Aventis Investigational Site Number 380001, Orbassano
  - Sanofi-Aventis Investigational Site Number 380002, Rozzano
- Spain (2):
  - Sanofi-Aventis Investigational Site Number 724001, Badalona
  - Sanofi-Aventis Investigational Site Number 724002, Barcelona
- United Kingdom (2):
  - Sanofi-Aventis Investigational Site Number 826001, Newcastle upon Tyne
  - Sanofi-Aventis Investigational Site Number 826002, Wolverhampton

REFERENCES:
- [Derived] Novello S, Besse B, Felip E, Barlesi F, Mazieres J, Zalcman G, von Pawel J, Reck M, Cappuzzo F, Ferry D, Carcereny E, Santoro A, Garcia-Ribas I, Scagliotti G, Soria JC. A phase II randomized study evaluating the addition of iniparib to gemcitabine plus cisplatin as first-line therapy for metastatic non-small-cell lung cancer. Ann Oncol. 2014 Nov;25(11):2156-2162. doi: 10.1093/annonc/mdu384. Epub 2014 Aug 19. PMID 25139550